CLINICAL TRIAL: NCT04054219
Title: Prospective, Single Center, Pivotal Investigation to Investigate Efficacy and Safety of WISHBONE HA, Used as Bone Graft Substitute for Different Indications Where Bone Grafting Procedures Are Required Before Implant Placement.
Brief Title: Evaluation of Efficacy and Safety of Wishbone HA as Bone Graft Substitute, a Pre-market Clinical Investigation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wishbone SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20181207_WHA_CIP
Record Dates: First submitted 2019-08-07; First posted 2019-08-13 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Bone Loss in Jaw

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Bone graft substitute — Evaluation of a device made of deproteinized bovine bone material as bone graft substitute in different indications requiring bone grafting procedures before implant placement

SUMMARY:
Evaluation of efficacy and safety of Wishbone HA as bone graft substitute, a pre-market clinical investigation.

Group1: Extraction Socket management Group 2: Sinus lift

ELIGIBILITY:
Inclusion Criteria:

* Subject signed the informed consent form
* Subject is ≥18 and ≤ 80 years old.
* Subject presented in need of:

  1. tooth extraction without estimated need of connective tissue grafting OR
  2. defect in the upper jaw requiring sinus lift with or without lateral augmentation procedure prior to implant placement
* The subject is willing and able to comply with all investigation related procedures (such as exercising oral hygiene and attending all follow-up visits).
* Full-mouth bleeding score (FMBS) lower than 25%
* Full-mouth plaque score (FMPI) lower than 25%
* The subject displays no clinical contraindications for a 2-stage surgical procedure

Exclusion Criteria:

* Less than 2 mm of remaining keratinized mucosa
* Severe vertical resorption of the crest (except internal resorptions, i.e. expanded sinuses)
* Ridge with prior bone augmentation procedure performed (i.e ridge preservation)
* Any disorders in the planned implant area such as previous tumors, chronic bone disease.
* Alcohol or drug abuse as noted in subject records or in subject history.
* Any ongoing application of interfering medication (steroid therapy, bisphosphonate, etc).
* Reason to believe that the treatment might have a negative effect on the subject's overall situation (psychiatric problems), as noted in subject records or history.
* Smoking: >10 cigarettes per day

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Measure of the bone augmentation success | 4 months after procedure
  Group 1 - Extraction Socket Management: Efficacy endpoint based on the bone augmentation success (bone gain after bone augmentation procedure) measured by Cone Beam CT
Measure of the bone augmentation success | 6 months after procedure
  Group 2 - Sinus lift: Efficacy endpoint based on the bone augmentation success (bone gain after bone augmentation procedure) measured by Cone Beam CT

SECONDARY OUTCOMES:
Safety endpoint: Collection of all device related adverse events | 4 months after procedure
  Group 1 - Extraction Socket Management: Collection of all device related adverse events reported by the investigator and by the patient from the time of procedure up to the time of implant insertion: Abnormal tissue reaction of the surrounding area, Not expected complications, Loss of material, Additional signs of Inflammation, Wound dehiscence, Membrane exposure, Persistent feeling of discomfort at the gingival incision
Safety endpoint: Collection of all device related adverse events | 6 months after procedure
  Group 2 - Sinus lift: Collection of all device related adverse events reported by the investigator and by the patient from the time of procedure up to the time of implant insertion: Abnormal tissue reaction of the surrounding area, Not expected complications, Loss of material, Additional signs of Inflammation, Wound dehiscence, Membrane exposure, Persistent feeling of discomfort at the gingival incision
Procedure success: ability to successfully perform the implants placement | 4 months after procedure
  Group 1 - Extraction Socket Management: The procedure is a success if the bone is sufficient for implant placement and implant can be placed successfully with sufficient good primary stability (>10Ncm) measured using a torque wrench.
Procedure success: ability to successfully perform the implants placement | 6 months after procedure
  Group 2 - Sinus lift: The procedure is a success if the bone is sufficient for implant placement and implant can be placed successfully with sufficient good primary stability (>10Ncm) measured using a torque wrench.
Site preparation: need for under or over preparation of the osteotomy | 4 months after procedure
  Group 1 - Extraction Socket Management: If the second CBCT shows favourable results, implant placement will be performed. Depending on the clinician's choice, a CAD-CAM surgical guide could be prepared to facilitate proper positioning of the implant(s). Access to the bone crest will be made with an as minimally-invasive surgical approach as possible, depending on the surgeon's choice.
  The drilling procedure will be performed according to the manufacturer's instructions for the placement the implant(s); during this drilling procedure, the clinician will determine if the bone quality is sufficient for placing the implant(s).
Site preparation: need for under or over preparation of the osteotomy | 6 months after procedure
  Group 2 - Sinus lift: If the second CBCT shows favourable results, implant placement will be performed. Depending on the clinician's choice, a CAD-CAM surgical guide could be prepared to facilitate proper positioning of the implant(s). Access to the bone crest will be made with an as minimally-invasive surgical approach as possible, depending on the surgeon's choice.
  The drilling procedure will be performed according to the manufacturer's instructions for the placement the implant(s); during this drilling procedure, the clinician will determine if the bone quality is sufficient for placing the implant(s).
Assessment of the bone quality and bone quantity | 4 months after procedure
  Group 1 - Extraction Socket Management: Bone quality and bone quantity will be assessed following Lekholm and Zarb classification.
Assessment of the bone quality and bone quantity | 6 months after procedure
  Group 2 - Sinus lift: Bone quality and bone quantity will be assessed following Lekholm and Zarb classification.
Implant survival | 1 year after after definitive prosthesis delivery
  Implant survival will be assessed by answering if:
  1. The implant remains in the jaw
  2. The implant is damaged to the extent that it cannot be restored
Implant success | 1 year after after definitive prosthesis delivery
  Implant Success will be defined in accordance with the criteria proposed by van Steenberghe. Answering yes or no to the following statements:
  1. The implant causes allergic, toxic or gross infectious reactions either locally or systemically.
  2. The implant offers anchorage to a functional prosthesis.
  3. The implant shows signs of fracture or bending.
  4. The implant shows signs of peri-implant radiolucency on an intra-oral radiograph using a paralleling technique strictly perpendicular to the implant-bone interface.
  5. The implant shows mobility when individually tested by tapping or rocking with a hand instrument.
Papilla index evaluation | 1 year after definitive prosthesis delivery
  The soft tissue contour adjacent to the implant is assessed from definitive prosthetic placement to the 1-year follow up visit using the papilla index according to Jemt 1997
Plaque index evaluation | 1 year after definitive prosthesis delivery
  The plaque accumulation is assessed using the modified Plaque Index (mPlI) according to Mombelli et.al:
  0 = No detectible plaque
  1 = Plaque only recognized by running a probe across the marginal surface of the implant 2 = Plaque can be seen by the naked eye 3 = Abundance of soft matter
Bleeding index evaluation | 1 year after definitive prosthesis delivery
  The bleeding tendency is assessed by a modified Sulcus Bleeding Index (mBI) according to Mombelli et. al:
  0 = No bleeding when a periodontal probe is passed along the gingival margin adjacent to the implant
  1. = Isolated bleeding spots visible
  2. = Blood forms a confluent red line on the margin 3 = Heavy or profuse bleeding
Keratinized mucosa evaluation | 1 year after definitive prosthesis delivery
  Classification will be performed as:
  0 = No keratinized mucosa around the implant.
  1= Keratinized mucosa Measurement in mm of the keratinized mucosa in the apico-coronal direction using a periodontal probe
Patient Oral health profile evaluation | 1 year follow-up visit
  The quality of life will be assessed at all visits by a questionnaire which is going to be completed be the subject. The shortened version from Brennan et al., OHIP-14 has been adopted for use in this investigation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium